CLINICAL TRIAL: NCT00848081
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design Study to Evaluate the Safety and Efficacy of Daily Tadalafil for 12 Weeks in Men With Signs and Symptoms of Benign Prostatic Hyperplasia on Concomitant Alpha1-Adrenergic Blocker Therapy
Brief Title: A Study of Tadalafil in Men With Benign Prostatic Hyperplasia Symptoms Who Are Being Treated With Alpha Blockers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief medical officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11668; H6D-MC-LVHS (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-08

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Prostate; BPH; Benign Prostatic Hyperplasia; BPH-LUTS; LUTS; Phosphodiesterase Inhibitors; tadalafil; alpha blockers
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Tadalafil (Experimental)
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — 5 mg taken by mouth once daily for 12 weeks
  Other Names: LY450190; Cialis
  Arms: Tadalafil
Drug: Placebo — By mouth once daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of tadalafil when given to men who are currently taking a medication called an alpha blocker for the treatment of benign prostatic hyperplasia (BPH) symptoms (such as urinary frequency, urgency, and a feeling that the bladder is not completely emptied after urination).

ELIGIBILITY:
Inclusion Criteria:

* Stable on alpha blocker therapy for the treatment of BPH for at least 4 weeks prior to starting the study.
* Have not taken the following treatments within the indicated duration and agree not to use at any time during the study:

  1. All other Benign Prostatic Hyperplasia therapy (including herbal preparations) for at least 4 weeks prior to receiving study medication.
  2. Overactive Bladder therapy (including antimuscarinics) for at least 4 weeks prior to receiving study medication.
  3. Erectile Dysfunction therapy (including herbal preparations) for at least 4 weeks prior to receiving study medication.
* If taking finasteride or dutasteride, must have been taking treatment for at least 6 months.

Exclusion Criteria:

* Currently receiving alpha-blocker therapy for the treatment of hypertension.
* History of symptoms associated with orthostasis, including recurrent episodes of dizziness, lightheadedness, loss of consciousness, or syncope.
* Treated with nitrates for any cardiac conditions.
* Have had any of the following in the past 90 days: Heart attack, also known as a myocardial infarction (MI); Heart bypass surgery (called coronary artery bypass graft surgery); Had a procedure to open up blood vessels in the heart known as angioplasty or stent placement (percutaneous coronary intervention).
* Have problems with kidneys, liver, or nervous system
* Have uncontrolled diabetes
* Have prostate cancer, are being treated for cancer or have clinical evidence of prostate cancer (PSA greater than 10 ng/ml at the start of study).
* Have had a stroke or a significant injury to brain or spinal cord.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM- 5 PM Eastern time (UTC/GMT -5 hourse, EST), Study Director — Eli Lilly and Company
Locations (31):
- United States (28):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anchorage, Alaska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paramount, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vacaville, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Clair Shores, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Missoula, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bay Shore, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden City, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poughkeepsie, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salisbury, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmond, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Menomonee Falls, Wisconsin
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo by mouth once daily for 12 weeks
- Tadalafil: Tadalafil 5 mg taken by mouth once daily for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Tadalafil
Started | 160 | 158
Completed | 140 | 140
Not Completed | 20 | 18
Not completed — Adverse Event | 6 | 7
Not completed — Protocol Violation | 8 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Total
Number analyzed (Participants) | 160 | 158 | 318
Age Continuous [Mean (Standard Deviation); unit: years] | 67.35 (9.13) | 67.41 (9.11) | 67.38 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 160 | 158 | 318
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 20 | 38
  Not Hispanic or Latino | 142 | 138 | 280
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — If a subject reported multiple race categories, he was counted as "more than one race" but not in any single category.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 14 | 17 | 31
    White | 144 | 137 | 281
    More than one race | 0 | 2 | 2
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 157 | 148 | 305
  Puerto Rico | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Men With Treatment-emergent Dizziness
Description: The primary safety measure is the proportion (reported in numbers) of subjects experiencing treatment-emergent dizziness to include the Medical Dictionary for Regulatory Activities (MedDRA) preferred terms of dizziness, dizziness postural, and procedural dizziness. Treatment-emergent dizziness is defined as any of the predefined terms of dizziness that is first reported or worsens in severity after baseline.
Time Frame: Baseline through 12 Weeks
Population: Primary Analysis Population-included all subjects who were randomized and took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 159 | 158
Participants | 9 | 11
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; The p-value is from a one-sided Fisher's exact test with a significance level of 0.05. A total of 142 subjects per treatment arm would provide 91% power to detect the difference between a Group 1 proportion of 0.03 and a Group 2 proportion of 0.13; Test type: Superiority or Other; p = 0.403, Fisher Exact — 1-sided test

2. Secondary Outcome: Number of Participants With Positive Orthostatic Vital Signs Test; Shift From Any Pre-Randomization to Any Post-Randomization Visit
Description: A positive orthostatic test is defined as at least one of the following 4 criteria being met at any pre-randomization or post-randomization visit: (1) reduction in systolic blood pressure of >= 20 mmHg from the supine to standing position;(2)reduction in diastolic blood pressure of >=10 mmHg from the supine to standing position;(3)increase in heart rate of >= 20 bpm from the supine to standing position; or (4)Unable to remain standing. A negative orthostatic test is defined as none of the above 4 criteria (1, 2, 3, or 4) being met at any pre-randomization or post-randomization visit.
Time Frame: Baseline through 12 Weeks
Population: All randomized subjects in the analysis population with non-missing data.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 158 | 156
Participants
  Positive Pre-Random. to Negative Post-Random. | 22 | 15
  Negative Pre-Random. to Positive Post-Random. | 21 | 19
  Positive Pre-Random. to Positive Post-Random. | 14 | 16
  Negative Pre-Random. to Negative Post-Random. | 101 | 106

3. Secondary Outcome: International Prostate Symptom Score (IPSS) Change From Baseline
Description: Change from baseline to endpoint in IPSS Score. The IPSS Total Score is obtained by combining the scores of the responses to 1 through 7 component questions. Each question is scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: Baseline, 12 Weeks
Population: Primary Analysis Population-included all subjects who were randomized and took at least one dose of study medication and had non-missing baseline and endpoint data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 156 | 156
units on a scale
  Baseline | 13.3 (6.57) [-2.01 to 0.26] | 13.87 (7.15) [-2.01 to 0.26]
  Change from Baseline | -1.49 (5.29) | -2.28 (5.65)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; The LS mean, standard error, 2-sided 95% confidence interval and p-value for the difference between placebo and tadalafil 5 mg are from an analysis of covariance (ANCOVA) model; Test type: Superiority or Other; p = 0.130, ANCOVA — p-value is on change from baseline

4. Secondary Outcome: Postvoid Residual Volume (PVR) Change From Baseline
Description: Change from baseline to endpoint in PVR volume. PVR is obtained by measuring with ultrasound the remaining urine in the bladder after urination.
Time Frame: Baseline, 12 Weeks
Population: All randomized subjects who had non-missing baseline and endpoint data.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 150 | 151
milliliters
  Baseline values | 70.7 (74.87) | 80.3 (80.78)
  Change from Baseline | -1.9 (82.86) | -8.1 (88.5)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.258, ANOVA — p-value is on change from baseline; The p-value is from Type III sums of squares ANOVA on rank-transformed data

5. Secondary Outcome: Uroflowmetry (Qmax) Change From Baseline
Description: Change from baseline to endpoint in Qmax. Qmax is defined as the peak urine flow rate (measured in milliliters per second [mL/second] using standard calibrated flowmeter).
Time Frame: Baseline, 12 Weeks
Population: All randomized subjects with non-missing data.
Measure: Mean (Standard Deviation); unit: milliliters per second
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 115 | 115
milliliters per second
  Baseline | 12.8 (5.88) | 11.8 (4.93)
  Change from Baseline | 0.6 (4.03) | 0.6 (3.67)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.828, ANOVA; P-value is from Type III sums of squares ANOVA on rank-transformed data; p-value is on change from baseline

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were collected from randomization until the subject completed the study.
Arm/Group | Placebo | Tadalafil
Serious Adverse Events (participants affected / at risk) | 3/160 | 2/158
Other Adverse Events (participants affected / at risk) | 53/160 | 65/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=160) | Tadalafil (N=158)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lead dislodgement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=160) | Tadalafil (N=158)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 2 (3)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 8 (9)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gingival disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Suprapubic pain (General disorders) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Whiplash injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 3 (3) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Oesophagogastroduodenoscopy (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 8 (10) | 10 (14)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (3) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 3 (4) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Testicular mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Colon polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin lesion excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days